CLINICAL TRIAL: NCT06170632
Title: Flare Type Self-expandable Metal Stents (SEMS) vs Plastic Stent for the Treatment of Difficult Common Bile Duct Stone: a Randomized Post-marketing Multicenter Italian Study
Brief Title: Flare Type Self-expandable Metal Stents (SEMS) vs Plastic Stent for the Treatment of Difficult Common Bile Duct Stone
Acronym: TEMASTI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, SILVIA COCCA, Principal investigator, Azienda Ospedaliero-Universitaria di Modena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12.2023
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Biliary Stones; Bile Duct Diseases; Bile Duct Obstruction
Keywords: Common bile duct lithiasis; Difficult lithiasis
MeSH Terms: conditions — Cholecystolithiasis; Bile Duct Diseases; Cholestasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): Intervention group (IG): Patients with flare type SEMS placement
  Interventions: Device: Biliary drainage
- Control group (CG) (Active Comparator): Control group (CG): Patients with plastic stent placement
  Interventions: Device: Biliary drainage

INTERVENTIONS:
Device: Biliary drainage — Biliary drainage with FC-SEMS Niti-S FLARE TYPE

SUMMARY:
Migration of stones from the gallbladder to the common bile duct (CBD) facilitated by gallbladder contractions can be listed as a complication of gallstones disease. In the case of common bile duct stone (CBDs) migration, an endoscopic cholangiopancreatography (ERCP) should be offered for both symptomatic and asymptomatic patients fit for the procedure. An ERCP with an adequate endoscopic sphincterotomy obtains a complete biliary clearance in about 80-90% of the patients[5]. Whilst most cases are successfully treated with such first-line approaches, about 10-15% need alternative and/or adjunctive techniques to achieve bile duct clearance. These conditions are generally defined as "difficult" bile duct stones, a broad category of cases that encompasses very different scenarios. In the case of irretrievable CBDs, the European Society of Gastrointestinal Endoscopy (ESGE) recommends the endoscopic placement of a temporary biliary plastic stent to warrant biliary drainage. Since their introduction, fully covered self-expanding metal stents (FCSEMS) have rapidly been adopted for the treatment of benign biliary conditions such as strictures, leaks, or bleeding. In a recent retrospective study it has been shown that FCSEMS are useful in the approach of difficult lithiasis of CBD with no significant adverse events associated. Moreover, a promising FC-SEMS with a particular prosthesis design (flare type - Niti-S "S-Type" Taewoong) could be even more useful since it reduces the frequent complication of fully covered stents which is the migration of the prosthesis. However, prospective data on the effectiveness and on the adverse events rate on the use of SEMS for incomplete stone CBDs clearance are still lacking. Therefore, the investigators aim to estimate the incidence of adverse events, complete biliary clearance, and migration rate after 3-6 month from ERCP index (stent positioning), comparing plastic stents vs FC-SEMS (Niti-S "flare type" - Taewoong).

DETAILED DESCRIPTION:
BACKGROUND

The presence of gallstones is a very common condition worldwide, especially in developed countries where it is estimated to affect 10-15% of the adult population and accounts for a great part of total gastrointestinal-related healthcare expenditures[1]. Fortunately, only 10-25% of gallstones became symptomatic in their lifetime with an annual incidence of 2-3% per year [2, 3]. Moreover, the worldwide increase in obesity and in the prevalence of non-alcoholic fatty liver disease (NAFLD) , which represents a risk factor for gallstones, could contribute to the rising gallstone disease prevalence[4]. Migration of stones from the gallbladder to the common bile duct (CBD) facilitated by gallbladder contractions can be listed as a complication of gallstones disease. In the case of common bile duct stone (CBDs) migration, an endoscopic cholangiopancreatography (ERCP) should be offered for both symptomatic and asymptomatic patients fit for the procedure[1, 3]. An ERCP with an adequate endoscopic sphincterotomy obtains a complete biliary clearance in about 80-90% of the patients[5]. Whilst most cases are successfully treated with such first-line approaches, about 10-15% need alternative and/or adjunctive techniques to achieve bile duct clearance[1, 5]. These conditions are generally defined as "difficult" bile duct stones, a broad category of cases that encompasses very different scenarios, including large or multiple stones, peculiar stone shapes (e.g., barrel-shaped), stones located above a stricture or impacted, intrahepatic stones, altered distal bile duct (oblique, narrowed, sigmoid-shaped). In the case of irretrievable CBDs, the European Society of Gastrointestinal Endoscopy (ESGE) recommends the endoscopic placement of a temporary biliary plastic stent to warrant biliary drainage[1, 5, 6].

Numerous non-randomized studies, both prospective and retrospective, showed that an indwelling plastic stent may reduce the number and the size of CBDs[7-9], although the mechanism by which the endoprosthesis contributes to the clearance of CBD is unclear. Probably, the continuous friction between the CBDs and the stent contributes to producing mechanical stress that facilitates the disruption of the stones[10]. Available data showed that the biliary plastic stent had a success rate ranging from 44 to 96% for stone removal after the previous ERCP[11-14]. Since their introduction, fully covered self-expanding metal stents (FCSEMS) have rapidly been adopted for the treatment of benign biliary conditions such as strictures, leaks, or bleeding. In a recent retrospective study it has been shown that FCSEMS are useful in the approach of difficult lithiasis of CBD with no significant adverse events associated[9]. However, comparative prospective data between plastic and metal stents are still lacking. Theoretically, FC-SEMS could be more effective compared to the plastic stent in producing stress forces that facilitate the stone disintegration, but the quality of this evidence is still very low due to lack of data.

Moreover, a promising FC-SEMS with a particular prosthesis design (flare type - Niti-S "S-Type" Taewoong) could be even more useful since it reduces the frequent complication of fully covered stents which is the migration of the prosthesis[15-17]. However, the majority of the data concerning SEMS migration rate are available for the treatment of benign biliary stricture, understandably, with a low rate of both distal and proximal migration[17]. However, prospective data on the effectiveness and on the adverse events rate on the use of SEMS for incomplete stone CBDs clearance are still lacking. A definitive biliary stenting is not recommended by ESGE guidelines, but it is warranted to completely remove the CBD stones during the second ERCP, if possible.

AIM The investigators aim to estimate the incidence of adverse events, complete biliary clearance, and migration rate after 3-6 month from ERCP index (stent positioning) comparing plastic stents vs FC-SEMS (Niti-S "flare type" - Taewoong).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 year-old with difficult common bile duct stones as defined by the current ESGE guidelines
* Patients with irretrievable biliary stone and incomplete biliary drainage

Exclusion Criteria:

* Biliary malignant obstruction
* Other type of biliary benign or malignant stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | 3 months
  To estimate the incidence of adverse events, complete biliary clearance, and migration rate after 3-6 month from ERCP index (stent positioning), comparing plastic stents vs FC-SEMS (Niti-S "flare type" - Taewoong).

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Modena - Endoscopy Department, Modena, MO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 1. Troncone E, Mossa M, De Vico P, Monteleone G, Del Vecchio Blanco G. Difficult Biliary Stones: A Comprehensive Review of New and Old Lithotripsy Techniques. Medicina (Mex). 2022;58:120. 2. Everhart JE, Khare M, Hill M, Maurer KR. Prevalence and ethnic differences in gallbladder disease in the United States. Gastroenterology. 1999;117:632-9. 3. Shabanzadeh DM. Incidence of gallstone disease and complications. Curr Opin Gastroenterol. 2018;34:81-9. 4. Gu S, Hu S, Wang S, Qi C, Shi C, Fan G. Bidirectional association between NAFLD and gallstone disease: a systematic review and meta-analysis of observational studies. Expert Rev Gastroenterol Hepatol. 2023;17:283-93. 5. Manes G, Paspatis G, Aabakken L, Anderloni A, Arvanitakis M, Ah-Soune P, et al. Endoscopic management of common bile duct stones: European Society of Gastrointestinal Endoscopy (ESGE) guideline. Endoscopy. 2019;51:472-91. 6. Dong S, Singh T, Zhao Q, Li J, Wang H. Sphincterotomy plus balloon dilation versus sphincterotomy alone for choledocholithiasis: a meta-analysis. 2019;51:763-71. 7. Katsinelos P, Kountouras J, Paroutoglou G, Chatzimavroudis G, Zavos C. Combination of endoprostheses and oral ursodeoxycholic acid or placebo in the treatment of difficult to extract common bile duct stones. Dig Liver Dis Off J Ital Soc Gastroenterol Ital Assoc Study Liver. 2008;40:453-9. 8. Lee TH, Han J-H, Kim HJ, Park SM, Park S-H, Kim S-J. Is the addition of choleretic agents in multiple double-pigtail biliary stents effective for difficult common bile duct stones in elderly patients? A prospective, multicenter study. Gastrointest Endosc. 2011;74:96-102. 9. Grande G, Pigò F, Avallone L, Bertani H, Mangiafico S, Russo S, et al. Is the use of fully covered metal stents effective in the treatment of difficult lithiasis of the common bile duct? Surg Endosc. 2022;36:5684-91. 10. Horiuchi A, Nakayama Y, Kajiyama M, Kato N, Kamijima T, Graham DY, et al. Biliary stenting in the management of large or multiple common bile duct stones. Gastrointest Endosc. 2010;71:1200-1203.e2. 11. Yang J, Peng J, Chen W. Endoscopic biliary stenting for irretrievable common bile duct stones: Indications, advantages, disadvantages, and follow-up results. Surg J R Coll Surg Edinb Irel. 2012;10:211-7. 12. Kochlef A, Gargouri D, Kilani A, Ouakaa A, Elloumi H, Kharrat J, et al. Retained common bile duct stones after endoscopic sphincterotomy: temporary and longterm treatment with biliary stenting. Tunis Med. 2011;89:342-6. 13. Jain SK, Stein R, Bhuva M, Goldberg MJ. Pigtail stents: an alternative in the treatment of difficult bile duct stones. Gastrointest Endosc. 2000;52:490-3. 14. Maxton DG, Tweedle DE, Martin DF. Retained common bile duct stones after endoscopic sphincterotomy: temporary and longterm treatment with biliary stenting. Gut. 1995;36:446-9. 15. Park DH, Lee SS, Lee TH, Ryu CH, Kim HJ, Seo D-W, et al. Anchoring flap versus flared end, fully covered self-expandable metal stents to prevent migration in patients with benign biliary strictures: a multicenter, prospective, comparative pilot study (with videos). Gastrointest Endosc. 2011;73:64-70. 16. Koksal AS, Eminler AT, Parlak E. Fully Covered Metal Stents Safely Facilitate Extraction of Difficult Bile Duct Stones. Surg Laparosc Endosc Percutan Tech. 2023;33:152-61. 17. Zheng X, Wu J, Sun B, Wu Y-C, Bo Z-Y, Wan W, et al. Clinical outcome of endoscopic covered metal stenting for resolution of benign biliary stricture: Systematic review and meta-analysis. Dig Endosc Off J Jpn Gastroenterol Endosc Soc. 2017;29:198-210. 18. Jang DK, Lee SH, Ahn DW, Paik WH, Lee JM, Lee JK, et al. Correction: Factors associated with complete clearance of difficult common bile duct stones after temporary biliary stenting followed by a second ERCP: a multicenter, retrospective, cohort study. Endoscopy. 2020;52:C4. 19. Jang DK, Lee SH, Ahn DW, Paik WH, Lee JM, Lee JK, et al. Factors associated with complete clearance of difficult common bile duct stones after temporary biliary stenting followed by a second ERCP: a multicenter, retrospective, cohort study. Endoscopy. 2020;52:462-8. 20. Hartery K, Lee CS, Doherty GA, Murray FE, Cullen G, Patchett SE, et al. Covered self-expanding metal stents for the management of common bile duct stones. Gastrointest Endosc. 2017;85:181-6.